CLINICAL TRIAL: NCT03288233
Title: Measurement of Exhaled Lower Respiratory Carbon Monoxide and Correlation With Previous Measures of Red Cell Lifespan
Brief Title: Exhaled Carbon Monoxide and Red Blood Cell Turnover
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cincinnati (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Principal Investigator, Robert Cohen, M.D., Professor of Medicine, University of Cincinnati
Other Study IDs: CR2_2015-1070
Record Dates: First submitted 2017-06-08; First posted 2017-09-20 (Actual); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Diabetes Mellitus; Healthy
Keywords: Hemoglobin A1c; HbA1c; End tidal carbon monoxide
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary Group
  Interventions: Diagnostic Test: Breath carbon monoxide measurement

INTERVENTIONS:
Diagnostic Test: Breath carbon monoxide measurement — Participants will be asked to breath in designed breathing circuits or hold their breath for short period of time and then their breath samples will be collected in special bags and the carbon monoxide and carbon dioxide will be measured with electrochemical techniques.

SUMMARY:
Hemoglobin A1C (HbA1c) is the cornerstone of blood sugar monitoring. As HbA1c is formed by the covalent reaction of glucose with hemoglobin throughout the lifespan of the red blood cell (RBC), it is used as a surrogate marker for integrated mean blood glucose over time. The HbA1c value therefore is dependent on the average amount of time the RBC spends in the circulation (mean RBC age or MRBC). However, our previous studies measuring red cell lifespan using either an age cohort label (ex vivo labeling with biotin) or a population label (stable isotope) have demonstrated, contrary to established dogma, that the MRBC varies substantially among individuals and is sufficiently variable to affect HA1c interpretation in a significant percentage of individuals with diabetes. Although the stable isotope method is suitable for clinical studies, it has limited potential for application to large population of subjects. A potential alternative to the stable isotope approach that could be applied routinely to the average patient in the clinic is measurement of exhaled carbon monoxide (eCO) concentration, a reflection of RBC heme turnover. In general, the primary advantage of applying exhaled breath analyses to human clinical diagnostics and therapeutic monitoring is that this technique is noninvasive, safe, simple, and provides near-real time measurements. The purpose of this observational study is to optimize the collection of eCO in a normal control population followed by measurement in a cohort of subjects previously assessed by either the SI or biotin methods for comparison.

DETAILED DESCRIPTION:
Recently Investigators have demonstrated that RBC lifespan has substantial inter-individual variation even in people without diabetes or obvious hematologic diseases affecting RBC lifespan (5,6). Investigators combined Endocrinology-Hematology research group has taken a leading role in applying state-of-the-art methods for RBC survival measurement.The published articles articles are now cited when investigators refer to the state of the art understanding of true RBC lifespan (7). Using a biotin labeling method that involves ex vivo labeling of cells with biotin and then re-infusion of those cells, Investigators were able to demonstrate that RBC lifespan is sufficiently heterogeneous even in the hematologically normal population with normal reticulocyte count to significantly affect HbA1c interpretation (5). Recognizing the limitations of the safe but relatively invasive biotin technique, Investigators more recently developed a stable isotope (SI) in which RBC heme is labeled with orally administered 15N-glycine (6). This is a benign and noninvasive technique and expands the scope of RBC lifespan studies to sizable epidemiologic and physiologic studies, a number of which investigators are initiating and planning.

However, the feasibility of making the findings translatable to widespread patient care has been perceived as a limitation to the merit of answering these scientific questions. The SI approach still requires multiple blood measurements over months (6). This proposed project is designed to test the feasibility of a method to satisfy the unmet clinical need for measuring RBC survival easily, noninvasively, and inexpensively. The goal is to access most individuals with or at risk for diagnosis of diabetes in or near most doctors' offices. Over the next year Investigators intend to determine whether exhaled alveolar carbon monoxide (eCO), a measure of heme breakdown and hence of RBC turnover, can be used in this manner to provide a single point measure of RBC lifespan. Interestingly, heme metabolism is the only known endogenous source of carbon monoxide in people (8) and there are recent studies by others suggesting its potential for measuring RBC lifespan (9,10) Now that technology has advanced to measure CO with sufficient sensitivity and cost, investigators will explore the use of instrumentation at the same time investigators expand their studies using the SI approach. The results from this method will be compared with a previous small population of subjects that had lifespan measured by biotin and/or SI technique.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be between age 18 and 75 years, non-pregnant, with a goal of equal gender and race (Caucasian vs. African-American) distribution

Exclusion Criteria:

* known hemoglobinopathy or RBC disorder
* positive pregnancy test (in women of child-bearing potential or are breast feeding or planning pregnancy during the course of the study;
* baseline serum creatinine >1.5 mg/dl
* CBC outside the normal range
* history of GI blood loss or coagulopathy
* urine microalbumin >100 mcg/mg creatinine (spot collection);
* transaminases >3 X the upper limit of normal
* presence of serum antibodies to biotinylated proteins (which could interfere with the biotin RBC labeling protocol)
* greater than or equal to NYHA stage 3 heart failure;
* active infection;
* known rheumatologic disease
* uncontrolled hypo-or hyperthyroidism or an underlying illness known to be associated with either body wasting or changes in serum proteins
* lung transplantation, irradiation, recent surgery, recent intensive care admission, asthma, COPD, cystic fibrosis, smoking, recent hematoma, uncontrolled hypo- or hyperthyroidism or an underlying illness known to be associated with either body wasting or changes in serum proteins (e.g. certain malignancies including multiple myeloma or tuberculosis).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults with Diabetes aged 18 to 75 years previously measured for red blood cell lifespan
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Average end expiratory alveolar concentration of Carbon monoxide (ppm) in morning before breakfast | four consecutive weeks
  In this preliminary phase of the study we use a device that has not been used in the United States before (Carbolyzer II, Taiyo, Japan) as a surrogate marker for red blood cell (RBC) removal or turnover in human subjects. Published studies and the company literature for the Carbolyzer mBA-2000 would suggest sufficient capability for the purposes of such measurements. This project will test more rigorously the validity of these specifications for this application. First, the detector will be standardized in more detail with measurement of the CO content of defined mixtures in the range needed for sufficient sensitivity. The device will calibrated prior with known concentrations of a mixture of carbon monoxide in air at three points (0-3-12 ppm). In addition, investigators will evaluate alternative CO detection devices for suitability which do not alter the experience of the participating subject or the accompanying risks and benefits.
Average end expiratory alveolar concentration of CO (ppm) in morning 30 min after breakfast | four consecutive weeks
  similar to outcome 1
Average end expiratory alveolar concentration of CO (ppm) 30 min after lunch | one day sampling
  similar to outcome 1
Average end expiratory alveolar concentration of CO (ppm) 5 hours after lunch | one day sampling
  similar to outcome 1

CONTACTS AND LOCATIONS:
Overall Officials: Robert Cohen, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share the IPD

REFERENCES:
- [Background] Khera PK, Smith EP, Lindsell CJ, Rogge MC, Haggerty S, Wagner DA, Palascak MB, Mehta S, Hibbert JM, Joiner CH, Franco RS, Cohen RM. Use of an oral stable isotope label to confirm variation in red blood cell mean age that influences HbA1c interpretation. Am J Hematol. 2015 Jan;90(1):50-55. doi: 10.1002/ajh.23866. PMID 25293624
- [Background] Coburn RF. The measurement of endogenous carbon monoxide production. J Appl Physiol (1985). 2012 Jun;112(11):1949-55. doi: 10.1152/japplphysiol.00174.2012. Epub 2012 Mar 22. PMID 22442030
- [Background] Strocchi A, Schwartz S, Ellefson M, Engel RR, Medina A, Levitt MD. A simple carbon monoxide breath test to estimate erythrocyte turnover. J Lab Clin Med. 1992 Sep;120(3):392-9. PMID 1517686